CLINICAL TRIAL: NCT07004088
Title: The Effect of Mandala Coloring on Symptom Burden and Self-Care in Female Dialysis Patients
Acronym: mandala and HD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Zehra Aydin, Assistant Professor, Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 29.05.2024/03.06.2024
Record Dates: First submitted 2025-05-17; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Dialysis; Symptoms; Self Care
Keywords: dialysis; symptom index; self care

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mandala group (Experimental): Female patients undergoing dialysis treatment in the dialysis unit were given mandalas for 20-30 minutes and asked to paint during 6 dialysis session, personal information form, "Dialysis Symptom Index Scale", "Self-Care Power Scale for Chronic Dialysis Patients" were filled before and after the sixth dialysis session, t
  Interventions: Behavioral: Mandala coloring
- Control Group (No Intervention): Female patients undergoing dialysis treatment in the dialysis unit were informed about the study. Volunteer consent form, personal information form, "Dialysis Symptom Index Scale", "Self-Care Power Scale for Chronic Dialysis Patients" were filled at the beginning and after the sixth dialysis session

INTERVENTIONS:
Behavioral: Mandala coloring — Female patients undergoing dialysis treatment in the dialysis unit were informed about the study. After women are informed about the effects of mandala application on health and how to paint mandala; voluntary consent form, personal information form, "Dialysis Symptom Index Scale", "Self-Care Power Scale for Chronic Dialysis Patients" were filled. One hour after the start of each dialysis session, the patients were given mandalas for 20-30 minutes and asked to paint. The women's own paints and mandalas were preserved for the next session. After the sixth dialysis session , the patients were asked to refill the scales with one-on-one interviews, and the verbal opinions and feedback of the patients about the application were taken.
  Arms: Mandala group

SUMMARY:
In kidney patients, especially the continuous dialysis treatment can cause symptoms which adversely affect patients' self-care abilities and quality of life. T Nonpharmacological methods can be used to reduce low and moderate symptoms. Mandala is one of the non-pharmacological approaches and is used in many areas with its therapeutic properties.

In the literature review on the effect of mandala application on dialysis patients symptoms and self care, no research was found. The aim of this study was to determine the effect of mandala coloring on dialysis symptoms and self-care of female patients receiving hemodialysis treatment.

Data were collected by using personal information form, Dialysis Symptom Index Scale, Self-Care Power Scale for Chronic Dialysis Patients.

As an intervention tool, a circular mandala and 12 felt paint were used in the study.

Study was designed as a randomized control study Intervention Group; voluntary consent form, personal information form, "Dialysis Symptom Index Scale", "Self-Care Power Scale for Chronic Dialysis Patients" were filled. One hour after the start of each dialysis session, the patients were given mandalas for 20-30 minutes and asked to paint. After the sixth dialysis session , the patients were asked to refill the scales with one-on-one interviews, and the verbal opinions and feedback of the patients about the application were taken.

Control Group; Female patients undergoing dialysis treatment in the dialysis unit were informed about the study. Volunteer consent form, personal information form, "Dialysis Symptom Index Scale", "Self-Care Power Scale for Chronic Dialysis Patients" were filled. After the sixth dialysis session, the women were asked to refill the scales.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older
* Able to communicate adequately
* No psychiatric problems
* No vision problems
* Receiving hemodialysis treatment for at least 6 months
* Willing and able to provide informed consent to participate in the study

Exclusion Criteria:

* Hemodialysis patients younger than 18 years of age
* Patients with physical or psychological limitations that interfere with -participation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 82 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
dialysis related symptom | After voluntary consent is obtained, the scale filled in by interviewing the patients one-on-one before the mandala painting attempt begins. 4 weeks after the completion of the mandala colouring the scale replenished
  Dialysis Symptom Index (DSI); The Dialysis Symptom Index (DSI) was developed by Weisbord et al. (2005) to determine the symptoms experienced by HD patients and the level of impact on patients. The Turkish reliability and validity of the scale was made by Önsöz and Yeşilbalkan (2013) and Cronbach's alpha value was reported as 0.84. DSI identifies 30 symptoms, either physical or emotional. In DSI, the symptoms experienced in the last week are answered as yes-no, and if the answer is yes, the extent to which the symptoms affected the patients who answered "yes" was evaluated as 0 = no, 1 = none, 2 = some, 3 = sometimes, 4 = very little, 5 = too much. The total scale score is obtained by adding the obtained scores. The score of the scale ranges from 0-150. The fact that the answers given to the scale increased towards 150 points indicates that the effect of the symptom in question increased. The internal consistency coefficient of the scale was determined as 0.84 (Usta, 2013).
Self-Care Agency Scale for Patients on Long-Term Dialysis | After voluntary consent is obtained, the scale filled in by interviewing the patients one-on-one before the mandala painting attempt begins. 4 weeks after the completion of the mandala colouring the scale replenished
  The scale was developed by Besey Ören in 2010 for HD and peritoneal dialysis patients. The Self-Care Agency Scale is an easily understandable, 22-item, 3-point Likert-type scale. The items are scored as follows: 0=I always apply, 1=I sometimes apply, and 2=I do not apply at all. It was created for people to express their status of applying selfcare habits in their daily lives. The patient is asked to choose the most appropriate option for him. The total score obtainable from the tool ranges between 0 and 44. Subscale scores are obtained by summing the item scores under each subscale. Accordingly, scores obtainable from the subscales are 0-12 for the use of medicine, 0-10 for diet, 0-8 for self-monitoring, 0-4 for hygienic care, and 0-6 for mental state. It shows that as the score obtained from the scale decreases, self-care ability decreases.16 The α coefficient of the scale was 0.67.

CONTACTS AND LOCATIONS:
Locations (1):
- Dialysis Center, Istanbul, Istanbul, Turkey (Türkiye)